CLINICAL TRIAL: NCT01141634
Title: A Pilot Trial of Homeopathic Treatment for Attention Deficit Hyperactivity Disorder in Children and Adolescents
Brief Title: A Pilot Trial of Homeopathic Treatment for Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: SickKids Foundation (Other); Centre for Addiction and Mental Health (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Heather Boon, Principal Investigator, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UToronto -25628; CAM09-213 (Other Grant/Funding Number: SickKids Foundation)
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder; ADHD; ADD; Homeopathy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Materia Medica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Homeopathic Remedies — Homeopathic remedies prepared according to the standards as set out by Health Canada

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a developmental disorder that presents during childhood, and is characterized by developmentally inappropriate levels of inattention and/or hyperactive-impulsive behavior. It is proposed that classical homeopathic treatment can reduce the symptoms of ADHD without serious side effects. This is an open label pilot feasibility study (36 participants). Participants, age 6-16, will consult with a homeopathic practitioner who will select treatments based on classical homeopathy principles. All participants will be assessed on a 4-weekly basis for a total of 36 weeks. The purpose of the study is to assess feasibility of recruitment and patient retention, to obtain pilot data on which to base a sample size calculation for future study, and to identify major safety concerns. The study will use single homeopathic medicines approved for over-the-counter use in Canada. The primary outcome measure will be the validated Conners 3rd Edition - Parent.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6-16 diagnosed with ADHD of any subtype according to DSM-IV criteria.
* Mentally competent participants able to adhere to the given protocol and treatments administered as interventions, and able to answer outcome measures.
* Primary caregiver (parent or guardian) has given informed consent; child participant gives ongoing assent throughout the study.

Exclusion Criteria:

* Changes to participants' medication for ADHD within 6 weeks of study onset.
* Diagnosis of additional mental health disorder including but not limited to: Conduct Disorder, Autism Spectrum Disorder, Bipolar Disorder, and Major Depressive Disorder. The patient should not have current suicidal or homicidal ideation.
* Participants should have no history of head injury of seizures, organ system damage and should have an estimated I.Q within the normal range.
* Pregnancy and Lactation

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Conners 3-Parent | 36 weeks

SECONDARY OUTCOMES:
MYMOP2 | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heather S Boon, PhD, Principal Investigator — University of Toronto
Locations (1):
- Riverdale Homeopathic Clinic, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Brule D, Sule L, Landau-Halpern B, Nastase V, Jain U, Vohra S, Boon H. An open-label pilot study of homeopathic treatment of attention deficit hyperactivity disorder in children and youth. Forsch Komplementmed. 2014;21(5):302-9. doi: 10.1159/000368137. Epub 2014 Sep 19. PMID 25427521